CLINICAL TRIAL: NCT02340416
Title: Tissue Oxygen Index and Pulsatility Index in Orthopedic Surgery: a NIRS and TCD Pilot Trial
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Clemens Kietaibl, M.D., Medical University of Vienna
Other Study IDs: 1633/2013
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Cerebral Microemboli
Keywords: orthopedic surgeries; general anesthesia
MeSH Terms: interventions — Ultrasonography, Doppler, Transcranial; Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: Transcranial Doppler Ultrasound, DWL Doppler BoxX
  Other Names: Near Infrared Spectroscopy, Hamamatsu Niro-200Nx

SUMMARY:
Cerebral microemboli (ME) are frequently generated during major orthopaedic surgery. The primary objective of this study was applying novel transcranial Doppler (TCD) ultrasound software algorithm to quantify (ME load/15 minutes) and qualify (particulate vs. gaseous) ME, detected as high-intensity transient signals (HITS) in both middle cerebral arteries (MCAs) before and after orthopaedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* hip prosthesis
* knee prosthesis
* shoulder prosthesis
* spine surgery

Exclusion Criteria:

* severe valvular heart defect
* acute neurological disorder

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: orthopedic patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Cerebral microemboli detection | prior and directly after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Anaesthesiology & Intensive Care, Vienna General Hospital, Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Kietaibl C, Engel A, Horvat Menih I, Huepfl M, Erdoes G, Kubista B, Ullrich R, Windhager R, Markstaller K, Klein KU. Detection and differentiation of cerebral microemboli in patients undergoing major orthopaedic surgery using transcranial Doppler ultrasound. Br J Anaesth. 2017 Mar 1;118(3):400-406. doi: 10.1093/bja/aex001. PMID 28199523